CLINICAL TRIAL: NCT02524522
Title: Perioperative Pulmonary Recruitment and Postoperative Monitoring of Integrated Pulmonary Index in Off-pump Coronary Bypass Grafting
Brief Title: Perioperative Mechanical Ventilation and Postoperative Monitoring of IPI
Acronym: WEAN-IPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Mikhail Y. Kirov, Professor, head of Anesthesiology dept., Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: WEAN-IPI
Record Dates: First submitted 2015-08-04; First posted 2015-08-14 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Mechanical Ventilation Complication; Postoperative Pulmonary Atelectasis
Keywords: Integrated Pulmonary Index; automated protocol-driven weaning; pulmonary recruitment maneuver
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- INTELLiVENT-ASV mode (Active Comparator): Active comparator: Discontinuation of mechanical ventilation in postoperative period will be provided using automatically driven mode - INTELLiVENT-ASV. In the INTELLiVENT-ASV mode target EtCO2 will be 30-35 mm Hg, target SpO2 - 94-98%, quick wean option - activated.
  Interventions: Device: INTELLiVENT-ASV mode
- SIMV mode (Active Comparator): Active comparator: Discontinuation from mechanical ventilation in postoperative period will be provided using physician driven protocol. The synchronized intermittent mandatory ventilation (SIMV) mode settings will be as follows: PEEP 5 cm of water, FiO2 to achieve SpO2 > 94 %. Inspiratory pressure will be adjusted to deliver a tidal volume (VT) of 8 mL/kg predicted body weight; pressure support will be 2 cm of water higher. Respiratory rate (RR) will be adjusted to provide EtCO2 of 30-35 mm Hg. Respiratory rate and inspiratory pressure will be decreased gradually every 30 minutes. After decrease of inspiratory pressure to 6 cm of water (8 cm of water in case of BMI > 30 kg/m2) and respiratory rate to 6/min, the spontaneous breathing trial (SBT) will be started.
  Interventions: Device: SIMV mode

INTERVENTIONS:
Device: INTELLiVENT-ASV mode — Discontinuation with INTELLiVENT-ASV mode: discontinuation from mechanical ventilation in the early postoperative period will be provided by quick-wean option of INTELLiVENT-ASV mode
  Arms: INTELLiVENT-ASV mode
Device: SIMV mode — Discontinuation with SIMV mode: discontinuation with SIMV mode: discontinuation from mechanical ventilation in the early postoperative period will be provided in SIMV mode using physician driven algorithm
  Arms: SIMV mode

SUMMARY:
This study evaluates the influence of alveolar recruitment maneuver, protocolized liberation from respiratory support and monitoring of Integrated Pulmonary Index on the duration of the mechanical ventilation and the number of pulmonary complications in the early postoperative period after cardiac surgery.

DETAILED DESCRIPTION:
The outcome of elective off-pump coronary artery bypass grafting (OPCAB) can be significantly compromised due to early postoperative pulmonary complications. The risk of pulmonary complications including acute respiratory distress syndrome (ARDS), atelectases, and early ventilator-associated pneumonia remains inappropriate. Therefore, the maneuvers improving pulmonary aeration and the early restoration of spontaneous breathing activity can be of clinical value. Protocol-driven liberation from mechanical ventilation (CMV) can decrease the duration of CMV as well as the number of pulmonary complications. INTELLiVENT-Assisted spontaneous ventilation (INTELLiVENT-ASV) is a new approach, that may be as effective as conventional protocol-driven liberation from CMV.

In parallel, the thorough postoperative monitoring of pulmonary function during both postoperative mechanical ventilation and spontaneous breathing is also of a great value. One of the novel approaches to respiratory monitoring is Integrated Pulmonary Index (IPI). The Integrated Pulmonary Index merges four vital parameters including end-tidal carbon dioxide (EtCO2), respiratory rate, pulse rate, and oxygen saturation (SpO2) measured by capnography and pulse oximetry into a single index value utilizing fuzzy logic model .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Elective OPCAB.

Exclusion Criteria:

* Participation in any other study.
* Morbid obesity (BWI > 40).
* The risk of pneumothorax after alveolar recruitment due to pulmonary emphysema.
* Constant atrial fibrillation with pulse rate exceeding 100/min.
* Inability to breathe easily through the nostrils and thus to gain good quality EtCO2 readings while breathing spontaneously, due to chronic rhinitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative mechanical ventilation | 24 hrs
  Participants will be followed for the duration of mechanical ventilation, an expected average of 4 hrs

SECONDARY OUTCOMES:
Reduced incidence of postoperative respiratory complications | up to 28 days postoperatively
  * Hypoxemia determined as partial pressure of oxygen in arterial blood/fraction of inspired oxygen (PaO2/FiO2) < 300 mm Hg.
  * Atelectases.
  * Nosocomial (ventilator-associated) pneumonia.
  * Hypoxemia determined as PaO2/FiO2 < 300 mm Hg.
  * Atelectases.
  * Nosocomial (ventilator-associated) pneumonia. Hypoxemia determined as PaO2/FiO2 < 300 mm Hg, atelectases, • Nosocomial (ventilator-associated) pneumonia.
Duration of intensive care unit stay | 72 hours
  Participants will be followed for the duration of the ICU stay, an expected average of 48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y KIrov, MD, PhD, Principal Investigator — Northern State Medical University
Locations (1):
- City hospital # 1 / Northern State Medical University,, Arkhangelsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Feasibility study on full closed-loop control ventilation (IntelliVent-ASV™) in ICU patients with acute respiratory failure: a prospective observational comparative study — http://www.ccforum.com/content/17/5/R196